CLINICAL TRIAL: NCT04493450
Title: NEMO - an App for Side Effect Management in Oncology
Acronym: NEMO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Thomas Seufferlein (Other)
Responsible Party: Sponsor-Investigator, Thomas Seufferlein, Professor, Head of Department, University of Ulm
Organization: University of Ulm (Other)
Other Study IDs: NEMO
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Cancer Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smartphone-users: Cancer patients who use smartphones
  Interventions: Other: Documentation of cancer treatment side effects

INTERVENTIONS:
Other: Documentation of cancer treatment side effects — Standardized documentation of occurred side effects

SUMMARY:
This study investigates the use of digital and standardized documentation by patients of frequently occurring adverse events in oncological therapies.

DETAILED DESCRIPTION:
This research study is structured as a Phase I and II clinical trial. In phase I, the feasibility of using a smartphone application to document adverse events that have occurred during oncological therapies by the patient will be investigated. In phase II we will investigate whether the use of the smartphone app allows an improvement of patient care by reducing occurred adverse events.

ELIGIBILITY:
Inclusion Criteria:

* infusional combination therapy with at least two chemotherapy substances with or without further targeted therapies
* combination of at least two immune-checkpoint inhibitors
* able to read and understand German

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded:

* severe neurological disorders
* severe psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Phase I:
  - 30 participants in total non-randomly divided into three age groups (< 55 years, 55-75 years, > 75 years) of 10 people each.
  Phase II:
  - 36 participants randomly assigned a group of 18 persons (smartphone users, non-smartphone users)
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Patient acceptance of a new medium of communication | 6 months
  Acceptance of documentation of occurring side effects of oncological therapies with new communication media
Phase II: Change of occurred adverse events | 6 months
  Changes of side effects by at least 1 degree according to CTCAE scoring in comparison to the study start

SECONDARY OUTCOMES:
Phase II: Doses of chemotherapy | 6 months
  Maintenance of chemotherapy doses through better adverse event management
Phase II: Incidence of adverse events | 6 months
  Incidence of treatment-emergent adverse events as assessed by the CTCAE scale

CONTACTS AND LOCATIONS:
Overall Officials: Seufferlein, Principal Investigator — University Hospital Ulm
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kestler AMR, Kuhlwein SD, Kraus JM, Schwab JD, Szekely R, Thiam P, Huhne R, Jahn N, Furstberger A, Ikonomi N, Balig J, Schuler R, Kuhn P, Steger F, Seufferlein T, Kestler HA. Digitalization of adverse event management in oncology to improve treatment outcome-A prospective study protocol. PLoS One. 2021 Jun 4;16(6):e0252493. doi: 10.1371/journal.pone.0252493. eCollection 2021. PMID 34086740